CLINICAL TRIAL: NCT02437474
Title: Impact of Elimination or Reduction of Dietary Animal Proteins on Cancer Progression and Survival - A Pilot Study
Status: Completed | Type: Observational
Sponsor: Rosa Aspalter (Other)
Collaborators: University Hospital Regensburg (Other)
Responsible Party: Sponsor-Investigator, Rosa Aspalter, Director of Research, Verein Essen und Krebs
Organization: Verein Essen und Krebs (Other)
Other Study IDs: EK-01
Record Dates: First submitted 2015-04-16; First posted 2015-05-07 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Neoplasms
Keywords: vegan diet; lacto-ovo-vegetarian diet; cancer; tumor remission
MeSH Terms: conditions — Neoplasms | interventions — Diet, Vegetarian; Diet, Vegan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Omnivorous diet: Participants are consuming meat, fish, milk/milk products, eggs, plant products.
  Interventions: Behavioral: Omnivorous diet
- Lacto-ovo-vegetarian diet: Participants are consuming milk/milk products, eggs, plant products but no meat, fish or by-products.
  Interventions: Behavioral: Lacto-ovo-vegetarian diet
- Vegan diet: Participants are consuming plant products but no meat, fish, milk/milk products, eggs or by-products as well as honey.
  Interventions: Behavioral: Vegan diet

INTERVENTIONS:
Behavioral: Omnivorous diet — Adopting or continuing the selected diet for 6 months (omnivorous)
  Groups: Omnivorous diet
Behavioral: Lacto-ovo-vegetarian diet — Adopting or continuing the selected diet for 6 months (lacto-ovo-vegetarian)
  Groups: Lacto-ovo-vegetarian diet
Behavioral: Vegan diet — Adopting or continuing the selected diet for 6 months (vegan)
  Groups: Vegan diet

SUMMARY:
The purposes of this study are

* to test the hypothesis that elimination or reduction of dietary animal proteins leads to an improved prognosis in tumor patients
* to estimate the effect size and thus to enable sample size calculations for further studies
* to test the feasibility and tolerance of different diets, especially a vegan diet, in cancer patients and to proof that a vegan diet does not lead to a deterioration of health, tumor progression or to malnutrition
* to test the online platform as a study platform
* to test validity of self reported and online generated data

DETAILED DESCRIPTION:
Participating cancer patients select one of 3 defined diets (omnivor/lacto-ovo-vegetarian/vegan) at baseline and will continue their prescribed oncological therapy at their attending physician/clinic.

Participants provide data (cancer history, tumor behavior, food frequency questionnaires, questionnaires referring to quality-of-life) at baseline and at 3 and 6 months with optional data entry points at 12 and 124 months and a follow up questionnaire at 12 and 24 months. Data is entered online via the study platforms www.essenundkrebs.net and www.foodandcancer.net in German and English language (no additional clinical visits are required).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Inclusion in a tumor treatment or follow-up program
* Age >18 years

Exclusion Criteria:

* Psychiatric treatment during the last 3 months
* Pregnancy
* Breast feeding
* BMI < 18,5 kg/m2
* Major difficulties with food intake (swallowing, lack of appetite) limiting food intake
* Participation in other studies requiring the attendance to a particular diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will be recruited in community via print media, internet and especially social media as well as referred by oncological clinics.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number / percentage of remissions | 6 months
  Percentages of remissions as defined be complete absence of a tumor - in an ITT (intention to treat) analysis

SECONDARY OUTCOMES:
Tumor diagnosis and tumor behaviour (complete remission / partial remission / no change / progression) | 3 and 6 months (optional: 12 and 24 months)
  In the fist questionnaire, tumor history (diagnosis, classification, stage, previous therapy) is entered. At months 0, 3, 6, 12 and 24 tumor stage at present time is asked again. Comparing the staging between time points, tumor behaviour is categorized into four groups: complete remission / partial remission / no change / tumor progression. This will be determined for each participant by two investigator independently.
Relapse-free interval | 0, 3, 6, 12 and 24 months
  A relapse is defined by a recurrence of a tumor after a tumor free interval.
Therapies, therapy tolerability and side-effects (vomiting, nausea, hair loss, weakness, diarrhea, polyneuropathy,...) | 0, 3 and 6 months (optional: 12 and 24 months)
  The study questionnaire contains questions referring frequently occuring symptoms in cancer patients and wether they are related to a certain therapy or to other factors. The option "others" is included in case the present symptoms are not covered by the listed symptoms.
Comorbidities | 0, 3 and 6 months (optional: 12 and 24 months)
  The study questionnaire contains questions referring frequently occuring diseases other than cancer and wether they are present now or were present in the past. The option "others" is included in case the present disease is not covered by the listed diseases.
Medication | 0, 3 and 6 months (optional: 12 and 24 months)
  The study questionnaire contains questions referring medications and supplements and the dosage.
Quality of life | 0, 3 and 6 months (optional: 12 and 24 months)
  The study questionnaire contains questions referring quality of live covering the Karnofsky Index, but additional dimensions, too (psychosocial wellbeing).
Acceptance and feasibility of the selected diet | 3 and 6 months (optional: 12 and 24 months)
  The study questionnaire contains questions referring ease and difficulties with the selected diet.
Dietary pattern | 0, 3, 6, 12 and 24 months
  The study questionnaire contains questions referring previous dietary patterns and the dietary pattern which will be followed for the time of study participation (6 months) as well as the reason for choosing the respective diet. There is a categorical question asking for dietary patterns as well a comprehensive food frequency questionnaire especially adopted for discrimination of plant an animal derived foods.
  In addition to the main study questionnaires, participants are asked to report any unplanned change in their diet during study participation.
Frequency, extent and duration of nutritional changes | 3 and 6 months (optional: 12 and 24 months)
  The results referring to nutrition and dietary patterns are evaluated in terms of change and duration of change in dietary patterns (in months).
Weight and nutritional status | 0, 3, 6, 12 and 24 months
  Weight is entered in kg and size in cm. BMI is calculated. Nutritional status is derived from weight changes, laboratory test results (albumin) and questions referring to eating problems contained in the study questionnaire.
Experience with / performance of study platform | 0, 3 and 6 months
  One question of the questionnaire asks for experience and usability of the comprehensive questionnaire in terms of content, understanding, effort und technical experience.
Validity checks for self reported data | 0, 3 and 6 months
  Several questions are repeated in the questionnaire in a slightly different way to check for consistency. Dietary patterns are checked via food frequency questionnaires and control questions in the laboratory test section.
Survival rates for end stages | 6 months, 12 and 24 months
  Survival rates are calculated from the participants still alive and dead. In case of a pending questionnaire a contact person is asked or a cancer registry checked (depending on the citizenship of the participant).

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Aspalter, MD, Study Director — Registered Association "Food and Cancer"
Locations (1):
- Verein Essen und Krebs, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Catany Ritter A, Egger AS, Machacek J, Aspalter R. Impact of Elimination or Reduction of Dietary Animal Proteins on Cancer Progression and Survival: Protocol of an Online Pilot Cohort Study. JMIR Res Protoc. 2016 Jul 29;5(3):e157. doi: 10.2196/resprot.5804. PMID 27473726